CLINICAL TRIAL: NCT04458753
Title: Effect of Lumbar Core Strengthening on Pain, Disability, Proprioception, and Quadriceps Strength in Knee Osteoarthritis
Brief Title: Effect of Lumbar Stabilization on Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Adel Motawea Elsayed Zedan, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/002731
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; Lumbar core strengthening exercises; Dpinal stabilization training
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Core Stability

STUDY DESIGN:
Intervention Model Description: Two groups; group A will be treated with exercises directed to lumbar and knee, group B will receive exercises directed to knee only. 3 sessions/ week for 4 weeks
Who Masked: Participant
Masking Description: Patients will not know in which group they assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar focused + knee focused exercise group (Experimental): Will receive strengthening of back , abdominal, and quadriceps muscles, and stretching if calf and Hamstring muscles
  Interventions: Other: Lumbar focused exercises; Other: Knee focused exercises
- Knee focused exercise group (Active Comparator): Will receive strengthening of quadriceps and stretching of calf and Hamstring muscles
  Interventions: Other: Knee focused exercises

INTERVENTIONS:
Other: Lumbar focused exercises — Transersus abdominis activation Multifidus activation Back extension exercise Curl up abdominal exercise
  Other Names: Core training; Core stability
  Arms: Lumbar focused + knee focused exercise group
Other: Knee focused exercises — Strengthening of quadriceps Stretching of calf and Hamstring muscles
  Other Names: Traditional knee program

SUMMARY:
This study will be conducted to investigate the role of lumbar core strengthening in reducing knee pain and disability, and improving knee proprioception and Quadriceps strength in patients with knee OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a highly prevalent degenerative joint disease that impacts quality of life and puts a burden on health care costs. Idiopathic knee OA is an age-related disease, with prevalence ranging from 19-28%. Aetiology of OA (whether systemic or mechanical) remains unclear.

Lumbar spine has been reported to be associated with knee joint because of the biomechanical interrelationship. Decreased lumbar lordosis (that may indicate weak back extensors) and range of motion (that may indicate weak core stabilizers) had significant correlations with an increased spinal inclination angle, which was an independent factor related to knee OA (by increasing knee flexion angle). Knee OA may radiate pain to the back that together lead to more limited hip motion causing overloaded knees. Convergence presents between nerve roots supplying mid-lumbar muscles and joints, and that supply femoral nerve and quadriceps. Progression of knee OA is associated with progression of lumbar spine osteoarthritis. Altered trunk kinematics may cause altered tibiofemoral kinematics.

Strengthening of trunk extensors may be very important for knee OA as fatiguing back extensors led to 1) increased quadriceps inhibition (QI) that may lead to poor attenuation of ground reaction forces and excessive forces on the knees, 2) altered standing postural control, 3) a forward-leaned posture that increases the external knee moments, 4) a reduction in trunk proprioception.

Core stabilization exercises combined with knee-focused exercise or combined with hip strengthening resulted in less pain and better function. Interestingly, these studies included only patellofemoral pain and OA patients. This program may benefit knee OA patients as well. Strength, neuromuscular training and lumbopelvic stabilization reduced muscle weakness (of quadriceps and hip abductors), pain, and disability in men with mild knee OA. However, specific role of lumbar core muscles on knee OA, their effect on wider population (including females) and their effect on higher severity knee OA are lacking.

Strengthening of trunk core muscles may help pelvic stability which found to be beneficial in improving the trunk and lower extremity movement control, hip muscles strength, gait speed and daily activities. However, this done in stroke patients, it is hypothesized to benefit knee OA patients as well. Assessment and treatment of the trunk musculature should be considered in the rehabilitation of patients who demonstrate abnormal lower-extremity kinematics as found in knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. Knee pain for most days of previous month
2. Age 40- 65 years Knee OA grade 2-3 on kellgren- Lawrence grading scale. Unilateral or bilateral (provided that they radiologically have one knee ≤ grade 1 on KL score, and clinically pain ≤2 in VAS. The more severally affected knee will be included in evaluation and treatment) BMI= 25-32 kg/m2.

Exclusion Criteria:

* Symptomatic hip OA Hip or pelvis trauma Knee or hip infection Congenital or developmental disorder of lower limbs Intra-articular corticosteroid or hyaluronic acid injection into the knee within the last 3 months.

Previous surgery of the affected knee or spine. Significant injury to the knee within the past 6 months. Any disease or medication worsens physical function or hampers with knee evaluation (e.g. rheumatoid arthritis, canal stenosis..).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Average Knee Pain during last week | 1year
  Measured with visual analogue scale; 10 cm line, zero: no pain, 10: worst pain, during last week
Quadriceps isometric strength | 1 year
  Measured with Hand held dynamometer from supine, knee flexed 30 degrees

SECONDARY OUTCOMES:
Disability | 1 year
  Measured with Aggregate locomotor function score ( sum if 3 timing scires; up and diwn 7 stairs, 8 m walk, rising from chair)
Knee Proprioception absolute angular error | 1year
  Active joint angular reproduction at 30 degree knee flexion from sitting using inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S Abdelsalam, Ass prof, Study Chair — Cairo University
Locations (1):
- Kasr AlAiny hospital, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Foroughi F, Sobhani S, Yoosefinejad AK, Motealleh A. Added Value of Isolated Core Postural Control Training on Knee Pain and Function in Women With Patellofemoral Pain Syndrome: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 Feb;100(2):220-229. doi: 10.1016/j.apmr.2018.08.180. Epub 2018 Sep 26. PMID 30267667